CLINICAL TRIAL: NCT03822182
Title: A Prospective Randomized Controlled Trial Examining the Effectiveness of a Single Shot of Liposomal Bupivicaine for Reducing Post-operative Pain and Narcotic Use in Outpatient Rotator Cuff Surgery
Brief Title: Single Shot Liposomal Bupivicaine in Rotator Cuff Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Brian Badman, Principal Investigator, Clinical Associate Professor, Department of Orthopedic Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1806933448
Record Dates: First submitted 2019-01-27; First posted 2019-01-30 (Actual); Results first posted 2020-09-01 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Rotator Cuff Tear; Pain, Postoperative
Keywords: liposomal bupivicaine; interscalene block
MeSH Terms: conditions — Rotator Cuff Injuries; Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: The medication administered in the interscalene block is the intervention in this study. There are three different types of interscalene blocks that will be administered in order to compare the independent effectiveness of LB with the effectiveness of LB plus dexamethasone. Study participants will be randomized into one of three groups. The treatment groups are listed below:
  Group 1 (Control) Group 2 Group 3 30 ml of 0.5% bupivacaine and 0.4ml. of dexamethasone 15ml 0.5% bupivacaine and 10ml of LB (Exparel) and 5.4ml normal saline 15ml 0.5% bupivacaine and 10ml LB (Exparel) and 0.4ml dexamethasone and 5ml normal saline
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blinded study, thus, neither the surgeon nor the patient will know which type of interscalene block is used. A total of 78 envelopes containing will be generated consisting of 26 with Group 1", 26 with "Group 2" and 26 with "Group 3" designation. Envelopes will be sealed and randomly chosen by the anesthesiologist prior to surgery. The anesthesiologist will randomly select one of the envelopes which will determine the treatment group and indicate medications that will be included in the interscalene block. Patients will be blinded to the medication utilized as well as the treating surgeon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control/Bupivicaine +DMSO (Other): Group 1 will serve as the control and receive the standard injection consisting 30 ml of 0.5% bupivacaine and 0.4ml (4 mg) of dexamethasone.
  Interventions: Drug: Dexamethasone
- Liposomal bupivicaine (Active Comparator): Group 2 will receive a block with 15ml 0.5% bupivacaine and 10ml (133mg) of liposomal bupivicaine (Exparel) and 5.4ml of Normal Saline
  Interventions: Drug: liposomal bupivicaine
- Liposomal Bupivicaine +DMSO (Active Comparator): Group 3 will receive 15ml of 0.5% bupivicaine and 10ml (133mg) of Liposomal Bupivicaine (Exparel) and 0.4ml (4mg) dexamethasone and 5ml normal saline
  Interventions: Drug: liposomal bupivicaine; Drug: Dexamethasone

INTERVENTIONS:
Drug: liposomal bupivicaine — The medication administered in the interscalene block is the intervention in this study. There are three different types of interscalene blocks that will be administered in order to compare the independent effectiveness of LB with the effectiveness of LB plus dexamethasone. Study participants will be randomized into one of three groups. The treatment groups are listed below:
  Group 1 (Control): 30 ml of 0.5% bupivacaine and 0.4ml (4 mg) of dexamethasone Group 2: 15ml 0.5% bupivacaine and 10ml (133mg) of LB (Exparel) and 5.4ml normal saline Group 3: 5ml 0.5% bupivacaine and 10ml LB (Exparel) and 0.4ml (4 mg) dexamethasone and 5ml normal saline
  Other Names: Exparel
  Arms: Liposomal Bupivicaine +DMSO; Liposomal bupivicaine
Drug: Dexamethasone — steroid that will be used in control as well as in group 3 to see if effect with liposomal bupivicaine is prolonged as has been shown with standard bupivicaine.
  Arms: Control/Bupivicaine +DMSO; Liposomal Bupivicaine +DMSO

SUMMARY:
This document is a protocol for a human research study. This study is to be conducted according to United States standards of Good Clinical Practice in accordance with applicable Federal regulations and institutional research policies and procedures.

Liposomal bupivacaine (LB) has been shown to decrease post-operative pain and narcotic use when administered perioperatively as a local injection during arthroplasty procedures. Studies have also demonstrated that LB used in conjunction with dexamethasone may increase the duration of effectiveness of LB. This study seeks to evaluate if there is a difference in post-operative pain and narcotic use when LB is administered in an interscalene block during outpatient rotator cuff repair surgery. Furthermore, this study aims to determine if the addition of dexamethasone with LB results in a prolonged decrease in post-operative pain and a reduction in narcotic use.

DETAILED DESCRIPTION:
Outpatient surgery has become the gold standard for arthroscopic rotator cuff repair. Innovations in pain management with regional anesthesia and multimodal techniques have greatly contributed to this transition over the past several decades. Despite overall improvements, uncontrolled postoperative pain leads to prolonged ambulatory stays, increased patient dissatisfaction, unexpected admissions to the hospital or visits to the Emergency Room after surgery, and a greater incidence of complications. Furthermore, in the wake of the "opioid epidemic", concerns with narcotic consumption and addiction have become heightened with regulations and laws recently enacted making prescribing and managing postoperative pain ever more difficult.

Interscalene nerve blockade for shoulder procedures has become an increasingly common technique to provide perioperative pain control with good efficacy, low complication rates and reduced narcotic consumption. While the utilization of ultrasound to help administer the block has aided in the accuracy providing a more consistent analgesic effect, its overall short duration (12-24 hours) remains one of the major limitations of this technique. Modalities to prolong its effect have included use of indwelling catheters and the addition of perineural dexamethasone.

Recently, liposomal bupivacaine (LB) (Exparel) was approved for single shot interscalene administration by the FDA. This medication has been purported to provide up to 72 hours of extended release of bupivacaine via its multivesicular and honeycomb-like structure that predictably breaks down resulting in a slow and sustained release of the medication.9 Although numerous studies have been conducted and several meta-analyses performed looking at the overall efficacy of local injections of LB for operative procedures in an inpatient setting, no study to date has independently assessed its efficacy in the new perineural indication for outpatient shoulder surgery. Furthermore, no study to date has compared the use of LB to the use of LB with dexamethasone in a perineural indication to see if the duration of efficacy is further prolonged with the addition of dexamethasone. All existing literature is in regard to use of liposomal bupivacaine injected locally within the surgical site. This will be the first study to examine the perineural use of LB for outpatient shoulder surgery, and to determine if there is a prolonged decrease in pain and a decrease in narcotic consumption with the use of LB with dexamethasone when delivered as an interscalene block in an ambulatory setting.

Utilizing a prospective randomized controlled trial, this study seeks to evaluate if there is a difference in post-operative pain and narcotic use when LB is administered in an interscalene block during outpatient rotator cuff repair surgery. Furthermore, this study aims to determine if the addition of dexamethasone with LB results in a prolonged decrease in post-operative pain and an overall reduction in narcotic use.

Primary Aims & Objective

Aim 1a: To determine if the use of LB in an interscalene block decreases patient-reported post-operative visual analogue pain scale (VAS) in patients undergoing outpatient rotator cuff surgery

Hypothesis: There will be a decrease in the visual analogue pain scale for up to 72 hours post-operatively among participants who receive LB or LB plus dexamethasone, as compared to the control group (bupivacaine plus dexamethasone).

Objective: Utilizing a prospective randomized controlled trial, post-operative patient-reported VAS pain (on a scale of 1-10) will be collected 3 times per day (every 8 hours) for 5 post-operative days (PODs), corresponding to a total of 120 hours after surgery. For each 24-hour period (corresponding to each POD), the pain scores will be averaged and compared between the three treatment groups (control, LB, and LB plus dexamethasone) for each of the 5 PODs.

Aim 1b: To determine if the use of LB plus dexamethasone in an interscalene block decreases patient-reported post-operative VAS pain for a longer duration than the LB or the control group (bupivacaine plus dexamethasone) in patients undergoing outpatient rotator cuff surgery

Hypothesis: There will be a decrease in visual analogue pain scale for greater than 72 hours post-operatively among participants who receive LB plus dexamethasone, as compared to the LB and the control group (bupivacaine plus dexamethasone).

Objective: Utilizing a prospective randomized controlled trial, post-operative patient-reported visual analogue pain scale (on a scale of 1-10) will be collected 3 times per day (every 8 hours) for 5 post-operative days (PODs), corresponding to a total of 120 hours after surgery. For each 24-hour period (corresponding to each POD), the pain scores will be averaged and compared between the three treatment groups (control, LB, and LB plus dexamethasone) for each of the 5 PODs.

Secondary Aims & Objectives

Aim 2a: To determine if there is a difference in time at which post-operative narcotics are first used among three groups receiving different interscalene blocks (LB plus dexamethasone, LB, and control) in patients undergoing outpatient rotator cuff surgery.

Hypothesis: Narcotic use will begin at a later time among those receiving LB plus dexamethasone, as compared to the LB and the control group (bupivacaine plus dexamethasone).

Objective: Utilizing a prospective randomized controlled trial, narcotic use will be collected at 8-hour increments for a total of 5 post-operative days (PODs), corresponding to a period of 120 hours post-surgery. The 8-hour time period during which a participant first begins using a narcotic will be recorded and compared between three treatment groups (control, LB, and LB plus dexamethasone).

Aim 2b: To determine if there is a difference in patient-reported post-operative narcotic use (measured in morphine equivalents) among three groups receiving different interscalene blocks (LB plus dexamethasone, LB, and control) in patients undergoing outpatient rotator cuff surgery.

Hypothesis: There will be a decrease in cumulative narcotic use (measured in morphine equivalents) among participants who receive LB plus dexamethasone, as compared to the LB and the control group (bupivacaine plus dexamethasone).

Objective: Utilizing a prospective randomized controlled trial, post-operative patient-reported narcotic use (measured by the number of tablets ingested and converted to morphine equivalents) will be collected 3 times per day at 8-hour increments for a total of 5 post-operative days (PODs), corresponding to a total of 120 hours after surgery. For each 24-hour period (corresponding to each POD), narcotic use will be tabulated and compared between three treatment groups (control, LB, and LB plus dexamethasone). Furthermore, cumulative narcotic use during the 5-day (120 hour) study period will be calculated and compared between three treatment groups (control, LB, and LB plus dexamethasone).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Primary diagnosis of rotator cuff tear
* Able to provide informed consent
* Is willing and able to accept text messages

Exclusion Criteria:

* Known allergies to the study medications.
* Known narcotic or alcohol abuse (< 3 months)
* Revision rotator cuff surgery
* Contraindication to regional anesthesia
* Current narcotic regimen or contract with pain management specialist
* Diagnosed with any of the following co-morbidities:

  * Pre-existing coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: brian badman, MD, Principal Investigator — Indiana University
Locations (1):
- American Health Network, Avon, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share

REFERENCES:
- [Background] Cao X, Pan F. Comparison of liposomal bupivacaine infiltration versus interscalene nerve block for pain control in total shoulder arthroplasty: A meta-analysis of randomized control trails. Medicine (Baltimore). 2017 Sep;96(39):e8079. doi: 10.1097/MD.0000000000008079. PMID 28953626
- [Background] Bramlett K, Onel E, Viscusi ER, Jones K. A randomized, double-blind, dose-ranging study comparing wound infiltration of DepoFoam bupivacaine, an extended-release liposomal bupivacaine, to bupivacaine HCl for postsurgical analgesia in total knee arthroplasty. Knee. 2012 Oct;19(5):530-6. doi: 10.1016/j.knee.2011.12.004. Epub 2012 Jan 28. PMID 22285545
- [Background] Surdam JW, Licini DJ, Baynes NT, Arce BR. The use of exparel (liposomal bupivacaine) to manage postoperative pain in unilateral total knee arthroplasty patients. J Arthroplasty. 2015 Feb;30(2):325-9. doi: 10.1016/j.arth.2014.09.004. Epub 2014 Sep 16. PMID 25282071

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was between November 2018 and January 2020 and inclusive of all patients with a torn rotator cuff in the clinical practice of the PI
Pre-assignment Details: A total of 78 patients were enrolled. 1 patient was excluded after inspect report showing current narcotic use. 1 patient was excluded for failure to submit data postoperatively.
Groups:
- Control/Bupivicaine+DMSO: Group 1 will serve as the control and receive the standard injection consisting 30 ml of 0.5% bupivacaine and 0.4ml (4 mg) of dexamethasone.
  Dexamethasone: steroid that will be used in control as well as in group 3 to see if effect with liposomal bupivicaine is prolonged as has been shown with standard bupivicaine.
- Liposomal Bupivicaine: Group 2 will receive a block with 15ml 0.5% bupivacaine and 10ml (133mg) of liposomal bupivicaine (Exparel) and 5.4ml of Normal Saline
  liposomal bupivicaine: The medication administered in the interscalene block is the intervention in this study.
- Liposomal Bupivicaine + DMSO: Group 3 will receive 15ml of 0.5% bupivicaine and 10ml (133mg) of Liposomal Bupivicaine (Exparel) and 0.4ml (4mg) dexamethasone and 5ml normal saline
  liposomal bupivicaine: The medication administered in the interscalene block is the intervention in this study.
Period: Overall Study
Arm/Group | Control/Bupivicaine+DMSO | Liposomal Bupivicaine | Liposomal Bupivicaine + DMSO
Started | 26 | 25 | 27
Completed | 26 | 24 | 26
Not Completed | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1 Control: Group 1 will serve as the control and receive the standard injection consisting 30 ml of 0.5% bupivacaine and 0.4ml (4 mg) of dexamethasone.
  Dexamethasone: steroid that will be used in control as well as in group 3 to see if effect with liposomal bupivicaine is prolonged as has been shown with standard bupivicaine.
- Group 2: Group 2 will receive a block with 15ml 0.5% bupivacaine and 10ml (133mg) of liposomal bupivicaine (Exparel) and 5.4ml of Normal Saline
  liposomal bupivicaine: The medication administered in the interscalene block is the intervention in this study. There are three different types of interscalene blocks that will be administered in order to compare the independent effectiveness of LB with the effectiveness of LB plus dexamethasone. Study participants will be randomized into one of three groups. The treatment groups are listed below:
- Group 3: Group 3 will receive 15ml of 0.5% bupivicaine and 10ml (133mg) of Liposomal Bupivicaine (Exparel) and 0.4ml (4mg) dexamethasone and 5ml normal saline
  liposomal bupivicaine: The medication administered in the interscalene block is the intervention in this study. There are three different types of interscalene blocks that will be administered in order to compare the independent effectiveness of LB with the effectiveness of LB plus dexamethasone. Study participants will be randomized into one of three groups. The treatment groups are listed below:
  Dexamethasone: steroid that will be used in control as well as in group 3 to see if effect with liposomal bupivicaine is prolonged as has been shown with standard bupivicaine.
- Total: Total of all reporting groups
Arm/Group | Group 1 Control | Group 2 | Group 3 | Total
Number analyzed (Participants) | 26 | 24 | 26 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 22 | 62
  >=65 years | 5 | 5 | 4 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 14 | 35
  Male | 15 | 14 | 12 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 26 | 76

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Postoperative Pain: VAS
Description: Patient-reported post-operative VAS pain (on a scale of 0-10 with zero implying no pain and 10 indicating severe pain), measured post operatively, in 8-hour increments, for a total of 96 hours post-surgery, Patients will be prompted via text message to provide VAS pain every 8 hours. If a response text message is not received, a phone call will be made to obtain the information. Patients who do not have a smart phone will receive a phone call or keep a personal log of VAS pain.
Time Frame: 4 days post procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Liposomal Bupivicaine: Group 2 will receive a block with 15ml 0.5% bupivacaine and 10ml (133mg) of liposomal bupivicaine (Exparel) and 5.4ml of Normal Saline
  liposomal bupivicaine: The medication administered in the interscalene block is the intervention in this study. There are three different types of interscalene blocks that will be administered in order to compare the independent effectiveness of LB with the effectiveness of LB plus dexamethasone. Study participants will be randomized into one of three groups. The treatment groups are listed below:
  Group 1 (Control): 30 ml of 0.5% bupivacaine and 0.4ml (4 mg) of dexamethasone Group 2: 15ml 0.5% bupivacaine and 10ml (133mg) of LB (Exparel) and 5.4ml normal saline Group 3: 5ml 0.5% bupivacaine and 10ml LB (Exparel) and 0.4ml (4 mg) dexamethasone and 5ml normal saline
- Liposomal Bupivicaine + DMSO: Group 3 will receive 15ml of 0.5% bupivicaine and 10ml (133mg) of Liposomal Bupivicaine (Exparel) and 0.4ml (4mg) dexamethasone and 5ml normal saline
  liposomal bupivicaine: The medication administered in the interscalene block is the intervention in this study. There are three different types of interscalene blocks that will be administered in order to compare the independent effectiveness of LB with the effectiveness of LB plus dexamethasone. Study participants will be randomized into one of three groups. The treatment groups are listed below:
  Group 1 (Control): 30 ml of 0.5% bupivacaine and 0.4ml (4 mg) of dexamethasone Group 2: 15ml 0.5% bupivacaine and 10ml (133mg) of LB (Exparel) and 5.4ml normal saline Group 3: 5ml 0.5% bupivacaine and 10ml LB (Exparel) and 0.4ml (4 mg) dexamethasone and 5ml normal saline
  Dexamethasone: steroid that will be used in control as well as in group 3 to see if effect with liposomal bupivicaine is prolonged as has been shown with standard
Arm/Group | Control/Bupivicaine+DMSO | Liposomal Bupivicaine | Liposomal Bupivicaine + DMSO
Number analyzed (Participants) | 26 | 24 | 26
units on a scale
  Postoperative day 1 VAS | 3.1 (1.9) | 3.5 (2.2) | 2.4 (1.8)
  Postoperative day 2 VAS | 3.3 (1.8) | 2.8 (2.0) | 2.8 (1.7)
  Postoperative day 3 VAS | 2.4 (1.6) | 3.2 (2.1) | 2.1 (1.3)
  Postoperative day 4 VAS | 1.9 (1.3) | 2.9 (1.9) | 2.3 (1.5)

2. Secondary Outcome: Patient Reported Post Operative Opioid Use
Description: Patient-reported post-operative opioid use (converted to morphine equivalents), collected post operatively, in 8-hour increments, for a total of 96 hours post-surgery Patients will be prompted via text message to provide the amount of narcotics (number of pills converted to morphine equivalents) taken over the course of the previous 8 hours. If a response text message is not received, a phone call will be made to obtain the information. Patients who do not have a smart phone will receive a phone call or keep a personal log of narcotic use.
Time Frame: 4 days post procedure
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Groups:
- Liposomal Bupivicaine + DMSO: Group 3 will receive 15ml of 0.5% bupivicaine and 10ml (133mg) of Liposomal Bupivicaine (Exparel) and 0.4ml (4mg) dexamethasone and 5ml normal saline
  There are three different types of interscalene blocks that will be administered in order to compare the independent effectiveness of LB with the effectiveness of LB plus dexamethasone. Study participants will be randomized into one of three groups. The treatment groups are listed below:
  Group 1 (Control): 30 ml of 0.5% bupivacaine and 0.4ml (4 mg) of dexamethasone Group 2: 15ml 0.5% bupivacaine and 10ml (133mg) of LB (Exparel) and 5.4ml normal saline Group 3: 5ml 0.5% bupivacaine and 10ml LB (Exparel) and 0.4ml (4 mg) dexamethasone and 5ml normal saline
  Dexamethasone: steroid that will be used in control as well as in group 3 to see if effect with liposomal bupivicaine is prolonged as has been shown with standard bupivicaine.
Arm/Group | Control/Bupivicaine+DMSO | Liposomal Bupivicaine | Liposomal Bupivicaine + DMSO
Number analyzed (Participants) | 26 | 24 | 26
morphine milligram equivalents
  POD 1 MME | 26.5 (22.0) | 22.8 (22.3) | 18.8 (12.8)
  POD 2 MME | 36.1 (22.9) | 21.9 (24.9) | 22.8 (17.7)
  POD 3 MME | 29.7 (24.9) | 17.8 (21.8) | 14.4 (14.7)
  POD 4 MME | 21.1 (17.9) | 18.1 (23.9) | 16.8 (16.2)

ADVERSE EVENTS:
Time Frame: 96 hours
Groups:
- Liposomal Bupivicaine + DMS): Group 3 will receive 15ml of 0.5% bupivicaine and 10ml (133mg) of Liposomal Bupivicaine (Exparel) and 0.4ml (4mg) dexamethasone and 5ml normal saline
  The treatment groups are listed below:
  Group 1 (Control): 30 ml of 0.5% bupivacaine and 0.4ml (4 mg) of dexamethasone Group 2: 15ml 0.5% bupivacaine and 10ml (133mg) of LB (Exparel) and 5.4ml normal saline Group 3: 5ml 0.5% bupivacaine and 10ml LB (Exparel) and 0.4ml (4 mg) dexamethasone and 5ml normal saline
  Dexamethasone: steroid that will be used in control as well as in group 3 to see if effect with liposomal bupivicaine is prolonged as has been shown with standard
Arm/Group | Control/Bupivicaine +DMSO | Liposomal Bupivicaine | Liposomal Bupivicaine + DMS)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT03822182/ICF_006.pdf
  • Study Protocol and Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT03822182/Prot_SAP_007.pdf